CLINICAL TRIAL: NCT06326736
Title: An Exploratory Clinical Study of Safety and Efficacy of Neoantigen mRNA Vaccines in the Treatment of Patients With Resectable Pancreatic Cancer
Brief Title: Study of Neoantigen mRNA Vaccines in Patients With Resectable Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: Jiangsu Synthgene Biotechnology Co.Ltd. (Unknown)
Responsible Party: Principal Investigator, Sizhen Wang, associate chief physician, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024NZKY-014-02
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
Keywords: mRNA vaccine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surgical Procedures, Operative; camrelizumab; Immune Checkpoint Inhibitors; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pancreatic Cancer (Experimental): Resectable primary pancreatic tumor
  Interventions: Procedure: Surgery; Drug: Camrelizumab; Biological: SJ-Neo006; Drug: Gemcitabine+Abraxane

INTERVENTIONS:
Procedure: Surgery — Tumors of patients with pancreatic cancer must be radiographically resectable, and subjects with histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1) will be selected for neoantigen vaccine creation.
  Other Names: Surgical resection
Drug: Camrelizumab — Camrelizumab will be administered 6 weeks post-tumor resection.
  Other Names: PD-1 inhibitor
Biological: SJ-Neo006 — SJ-Neo006 will be prepared as personalized tumor Vaccines and administered 9 weeks post-tumor resection (+/- 2 weeks).
  Other Names: Neoantigen mRNA Vaccines
Drug: Gemcitabine+Abraxane — Gemcitabine+Abraxane regimen will be administered 21 weeks post-tumor resection.
  Other Names: chemotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of treating pancreatic cancer with surgery to remove cancerour tissue, followed by camrelizumab and a personalized cancer mRNA vaccines.

DETAILED DESCRIPTION:
The first purpose of this study is to evaluate the safety of treating pancreatic cancer with surgery to remove cancerour tissue.

Following with camrelizumab and a personalized Neoantigen mRNA Vaccines, and then with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this clinical study and sign the Informed Consent Form (ICF).
* Subjects must be >/= 18 years of age at time of informed consent.
* Subjective with radiographically resectable primary pancreatic tumors with radiographic features consistent with adenocarcinoma will be evaluated for surgical resection.
* Subjects with histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1) will be selected for neoantigen vaccine creation.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group (ECOG).
* Subjects must not have had prior chemotherapy, radiation therapy, or immunotherapy for Pancreatic ductal adenocarcinoma（PDAC）.
* Subjects with estimated survival > 12 weeks.

Exclusion Criteria:

* Prior neoadjuvant treatment, radiation therapy, anti-PD-1 antibody or any other immune therapy for pancreatic ductal adenocarcinoma.
* Known hypersensitivity or allergy to the active substance or to any of the excipients of SJ-neo006, Camrelizumab, Gemcitabine, Abraxane.
* Actie, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.
* Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection or subjects receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the investigator, increase the risk of serious neutropenic complications.
* Pregnancy, breastfeeding, or intending to become pregnant during the study or within 90 days after the last dose of study treatment.
* New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysthythmia, or electrocardiogram abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder.
* History or autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease.
* Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 2 years
  To observe and evaluate the safety of Neoantigen mRNA vaccine combined with Camrelizumab, for the number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 3,6,12 months
  The efficacy of Neoantigen mRNA vaccine combined with Camrelizumab by tumor lesion recurrence cycle at different time.

CONTACTS AND LOCATIONS:
Overall Officials: Xinbo Wang, MD, Study Director — Jinling Hospital, China
Locations (1):
- Wang Sizhen, Nanjing, Jiangsu, China